CLINICAL TRIAL: NCT06896955
Title: Effects of Virtual Reality Application and Progressive Relaxation Exercise Training on Pregnant Women's Stress, Birth Affect and Birth Self-Efficacy
Brief Title: Effects of Virtual Reality Application and Progressive Relaxation Exercise
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Sule Gokyildiz Surucu, Sule Gokyildiz Surucu, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 01.09.2023/55
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Pregnancy; Exercise; Virtual Reality
Keywords: Pregnancy; Exercise; progressive exercise; virtual reality
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PMR Group (Experimental): * After meeting the pregnant woman in the polyclinic, a personal information form and the Pregnancy Stress Assessment Scale will be filled out at the beginning of the research.
  * PMR will be explained to the pregnant woman and the first application will be done together. Any questions the pregnant woman may have will be answered.
  * An education booklet will be given about PMR.
  * The application will be performed 3 times a week starting at the 32nd week of pregnancy until labor begins, each application lasting 20 minutes.
  * The first application will be done face to face, and subsequent applications will be done by the pregnant woman herself, accompanied by a PMRvideo.
  * Continuous communication will be maintained with the pregnant woman via mobile phone.
  * The Pregnancy Stress Assessment Scale will be filled out at the 38th week.
  * The Birth Affect Scale and Birth Self-Efficacy Scale will be filled out on the first day after birth.
  Interventions: Other: PMR Education
- VR+PMR Group (Experimental): * PMR will be applied to this group accompanied by a therapeutic video shown with virtual reality glasses.
  * At the beginning of the research, a personal information form and the Pregnancy Stress Assessment Scale will be filled out.
  * An educational booklet about PMR will be given.
  * After both application methods are shown and applied, PGE will be applied together accompanied by a therapeutic video shown with virtual reality glasses.
  * The application will be performed 3 times a week starting from the 32nd week of pregnancy until labor begins, 20 minutes each time.
  * The first application will be done face to face, and subsequent applications will be done by the pregnant woman herself.
  * Pregnancy Stress Assessment Scale will be filled out again in the 38th week.
  * On the first day after delivery, the Birth Affect Scale, Birth Self-Efficacy Scale and Virtual Reality Glasses Application Evaluation Form will be filled out.
  Interventions: Other: PMR+VR Education
- Control Group (No Intervention): * Pregnant women in the control group will not be subjected to any treatment other than routine pregnancy follow-up and examinations at the hospital.
  * Forms will be filled out in parallel with the intervention groups.
  * Participants who wish will be given an educational booklet about PGE at the end of the study.

INTERVENTIONS:
Other: PMR+VR Education — PMR and VR education
  Arms: VR+PMR Group
Other: PMR Education — PMR education
  Arms: PMR Group

SUMMARY:
In the study, random assignment and randomization concealment will be applied to control selection bias. Pregnant women were assigned to groups by an independent statistician using the block randomization method. For this purpose, 6-digit combinations consisting of the letters "A", "B" and "C" were first created in the randomization of 78 women.

DETAILED DESCRIPTION:
There will be three groups in the randomized experimental controlled study:PRE (Progressive Relaxation Exercise), VR (Virtual Reality)+PGR (Progressive Relaxation Exercise) and Control group. In order to carry out the application phase of the study, the responsible researcher participated in the training program on PRE and received a certificate on this subject. In addition, permission for the use of PRE Cd was obtained from the Turkish Psychologists Association to be used in the PRE group. The following procedures will be performed for pregnant women included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation
* No communication difficulties (no mental retardation, no visual/hearing impairment)
* Knowing Turkish and being literate
* No fetal anomalies
* Being in the 32nd week of pregnancy
* Not being diagnosed with a risky pregnancy (multiple pregnancy, premature rupture of membranes, preeclampsia, gestational diabetes, placenta previa, etc., pregnancies may end with a cesarean section)

Exclusion Criteria:

* Having a psychiatric disease diagnosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-03-25 (Estimated); Primary Completion 2025-08-25 (Estimated); Study Completion 2026-03-25 (Estimated)

PRIMARY OUTCOMES:
Pregnancy Stress Assessment Scale | pre-intervention, after 2 month
  Change in pregnancy-related stress levels in pregnant women. As the score from the scale increases, stress increases.
Birth Self-Efficacy Scale | intervention after 2 month
  Change in self-efficacy levels of pregnant women during labor. As the score from the scale increases, self-efficacy increases.
Birth Affect Scale | intervention after 2 month
  Change in the emotional state experienced by mothers during labor. As the score from the scale increases, positive affect increases.

CONTACTS AND LOCATIONS:
Overall Officials: Senay Dagilgan, Msc, Principal Investigator — Cukurova University
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No